CLINICAL TRIAL: NCT01361191
Title: Early Treatment Stratification Based on PET Scan Response to R-MEGACHOP Followed by R-MEGACHOP or R-IFE Plus Peripheral Autologous Stem Cell Transplant (PBSCT) in Patients With Poor Prognosis DLBCL
Brief Title: Early Treatment Stratification Based on PET Scan Response to Chemotherapy in Patients With Diffuse Large B-cell Lymphoma
Acronym: R-MEGACHOP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEL/TAMO-2006; EudraCT number 2006-005254-68
Record Dates: First submitted 2008-04-14; First posted 2011-05-26 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Diffuse Large B-cell Lymphoma; Follicular Grade 3B Lymphoma
Keywords: DLBCL; PET; IPI; R-MegaCHOP; Autologous stem cell transplantation
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: R-MEGACHOP — * If PET + after third cycle: 2 cycles of R-IFE followed by PBSCT
  * If PET - after third cycle: 3 additional cycles of R-MegaCHOP - R-MegaCHOP: cycles every 21 days RITUXIMAB Dosage: 375mg/m2, IV, day 1 CICLOPHOSPHAMIDE Dosage: 1500 mg/m2, IV, day 1 DOXORUBICIN Dosage: 65 mg/m2, IV, day 1 VINCRISTIN: Dosage 1.4 mg/m2 (max. 2.0 mg/m2, IV, day 1 PREDNISONE Dosage: 60 mg/m2, IV, day 1-5
  R-IFE: 2 cycles every 21 days:
  IFOSFAMIDE Dosage: continuous perfusion of 10 gr/m2/iv during 72 hours. Therefore, 3.33 gr/m2/corporal weight 24 hours day +1, +2 and +3.
  ETOPOSIDE Dosage: total 900 mg/m2, IV, which is 150 mg/m2 during 12 hours (days +1, +2 and +3).

SUMMARY:
The aim of the study is to evaluate the event free survival at three years in patients with diffuse large B-cell lymphoma with poor prognostic factors receiving R-MegaCHOP as induction therapy. Patients with positive PET after three cycles of R-MegaCHOP receive early salvage treatment with R-IFE and autologous stem cell transplantation. Patients with negative PET after three cycles of R-MegaCHOP are treated with three additional cycles of R-MegaCHOP without transplant.

DETAILED DESCRIPTION:
In addition to the above:

* To evaluate the overall survival after three years.
* To determine the rate of global responses and complete remissions, uncertain and partial.
* To determine the duration of the complete response after the treatment termination.
* To carry out an exploratory follow up of the event free survival and the overall survival at 5 years.
* To evaluate the treatment toxicity according CTC criteria (version 3.0) of the National Cancer Institute (NCI).
* To asses the role of PET in the disease stage and response evaluation compared to CAT.
* To identify the predictable response factors after 6 cycles of treatment with R-MegaCHOP administrated every 21 days; or 3 cycles of R-MegaCHOP, followed by IFE+TAPH in patients with DLBCL of severe prognosis.
* To evaluate the therapeutic fulfillment of the R-MegaCHOP and R+IFE cycles of treatment and/or R-IFE in reference with delays with the cycles administration and reductions of the chemotherapy dose (planned dose administrated in the planned term).

ELIGIBILITY:
Inclusion Criteria:

1. follicular lymphoma grade III diagnosed patients, diffuse large B-cell lymphoma, histologically confirmed with CD20+
2. aged between 18 and 65 years. Patients aged from 65 to 70 years can be included according to the investigator's criteria regarding the patients' global health status and the absence of excluding comorbidity.
3. IPI adjusted to the age over 1 or a-IPI and beta2-microglobulin equal or higher than 3 mg/dl 3. Punctuation in the ECOG grade from 0 to 4
4. Life expectancy over 12 weeks
5. Written informed consent form 6. New diagnosed patient without any previous treatment

Exclusion Criteria:

1. Existence of severe cardiac, pulmonary, neurologic, psychiatric and metabolic diseases not caused by the lymphoma.
2. uncontrolled high blood pressure (diastolic pressure in rest > 115 mmHg)
3. Altered hepatic function (bilirubin or AST/ALT superior or equal at 2 times the superior limit of normality) or renal (creatinine equal or superior at 1.5 times the superior limit of normality) not caused by the lymphoma.
4. other malignant neoplasias along the past 5 years, except skin tumors, excluded melanoma or carcinoma in situ of cervix
5. patients positive for HIV
6. patients with transformed follicular lymphoma
7. pregnant women or in nursing; women of childbearing age who do not use an adequate contraceptive method before being included in the study
8. ventricular ejection fraction inferior to 50%
9. patients with severe psychiatric diseases which can interfere with their ability for understanding the study (including alcoholism or drug addiction)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2007-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Event free survival at 3y in pat with DLBCL with a-IPI>1 or a-IPI=1 and ß2 µglobulin>=3mg/dl in pat PET+ after 3cycles of R-MegaCHOP and early rescue with R-IFE+TAPH or in pat PET- after 3cycles R-MegaCHOP followed by 3cycles of R-MegaCHOP without TAPH | 5 years follow-up

SECONDARY OUTCOMES:
To evaluate the overall survival after three years. Further secondary outcomes as described in study summary. | 5 years follow-up

CONTACTS AND LOCATIONS:
Overall Officials: José Fuster, MD, Principal Investigator — Son Dureta Hospital; Carlos Grande, MD, Principal Investigator — 12 Octubre Hospital; José Luís Bello, MD, Principal Investigator — Santiago Hospital; Maria José Ramirez, MD, Principal Investigator — Jerez Hospital; Carlos Panizo, MD, Principal Investigator — Navarra Clinic; Elena Pérez, MD, Principal Investigator — Morales i Meseguer Hospital; Jorge Gayoso, MD, Principal Investigator — Gregorio Marañon Hospital; Reyes Arranz, MD, Principal Investigator — Princesa Hospital; Eulogio Conde, MD, Principal Investigator — Marques de Valdecilla Hospital; Eva González, MD, Principal Investigator — Duran i Reynals Hospital; Miguel Canales, MD, Principal Investigator — La Paz Hospital; Joan Bargay, MD, Principal Investigator — Son Llatzer Hospital; Miguel T. Hernández, MD, Principal Investigator — Canarias University Hospital; Antonio Alcala, MD, Principal Investigator — Jaen Hospital; Luis Palomera, MD, Principal Investigator — Lozano Blesa Clinic; José Queizán, MD, Principal Investigator — Segovia Hospital; María José Peñarrubia, MD, Principal Investigator — Río Hortega Hospital; Alejandro Martín, MD, Principal Investigator — Virgen de la Concha Hospital; Sílvia Fernández, MD, Principal Investigator — León Hospital
Locations (19):
- Spain (19):
  - ICO- Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital de Jerez, Jerez de la Frontera, Cádiz
  - Hospital Clínico Univ. de Santiago, Santiago de Compostela, Galicia
  - Complejo Hospitalario de Jaén, Jaén, Jaén
  - Hospital Universitario La Princesa, Madrid, Madrid
  - Hospital Universitario Gregorio Marañon, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Univ. Son Dureta, Palma de Mallorca, Mallorca
  - Hospital Son Llàtzer, Palma de Mallorca, Mallorca
  - Hospital Univ. Morales Meseguer, Murcia, Murcia
  - Clínica Universitaria de Navarra, Pamplona, Pamplona
  - Hospital Universitario de Salamanca, Salamanca, Salamanca
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz de Tenerife
  - Hospital General de Segovia, Segovia, Segovia
  - Hospital Universitario Río Hortega, Valladolid, Valladolid
  - Hospital Universitario Virgen de la Concha, Zamora, Zamora
  - Hospital Clínico Lozano Blesa, Zaragoza, Zaragoza